CLINICAL TRIAL: NCT01429675
Title: Randomized, Open-label Crossover Study to Evaluate Comparative Pharmacokinetics of Ibandronate Between DP-R206(150mg Ibandronate / 24,000 IU Vitamin D3 Complex Tablet) and a 150mg Ibandronate Tablet in Healthy Adult Volunteers
Brief Title: Safety and Pharmacokinetic Characteristics of DP-R206 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DP-CTR206-01
Record Dates: First submitted 2011-08-23; First posted 2011-09-07 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2011-09

CONDITIONS: Healthy
MeSH Terms: interventions — Ibandronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bonviva (Active Comparator)
  Interventions: Drug: bonviva
- DP-R206 (Experimental)
  Interventions: Drug: bonviva

INTERVENTIONS:
Drug: bonviva — 150mg Ibandronate once a month
  Other Names: DP-R206 : DP11012; bonviva : B1184B01

SUMMARY:
The purpose of this study is compare the pharmacokinetic characteristics of DP-R206 (150mg Ibandronate / 24,000 IU Vitamin D3 complex tablet, qd) and Bonviva (150mg Ibandronate, qd) after oral administration in healthy adult volunteers.

DETAILED DESCRIPTION:
The number of patient is eighty-four. Patients were randomly assigned either a Bonviva tablet(150mg Ibandronate, qd) first, DP-R206(150mg Ibandronate / 24,000 IU Vitamin D3 complex tablet, qd) Second or DP-R206(150mg Ibandronate / 24,000 IU Vitamin D3 complex tablet, qd) first, Bonviva tablet(150mg Ibandronate, qd) second.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 55 years of healthy volunteers

Exclusion Criteria:

* Hypersensitivity Reaction about Ibandronate or other drugs(aspirin, antibiotics)

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetics | predose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 24, 32, 48, 72, 120 hours post-dose
  Cmax, AUClast

SECONDARY OUTCOMES:
Composite of pharmacokinetics | predose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 24, 32, 48, 72, 120 hours post-dose
  AUCinf, tmax, t½β

CONTACTS AND LOCATIONS:
Overall Officials: Kyun seop Bae, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea